CLINICAL TRIAL: NCT00925964
Title: Interest of Measuring the Systolic Pressure Index in Assessing the Risk of Cardiovascular Events Peri-operatively in the Surgery, Settled Out of Cardiovascular Surgery
Brief Title: Systolic Pressure Index in Assessing the Risk of Cardiovascular Events
Acronym: IPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I07029
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2009-06

CONDITIONS: Cardio-vascular Events

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample to evaluate Troponin, a Cardiac biomarker
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients exposed: Patients with Systolic Pressure Index <0,9 ou >1,4.
- Patients not exposed: Patients with Systolic Pressure Index >0,9 ou <1,4.

SUMMARY:
To investigate whether the presence of a Systolic pressure index (<0.9 or> 1.4) is a marker of risk of cardiovascular events after peri-operative high-risk surgery outside the cardiac and vascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* age> 40 years
* surgery set :
* Visceral surgery: gastrectomy or colectomy, abdomino-perineal amputation, pancreatic surgery, liver surgery, esophageal surgery
* In urological surgery: nephrectomy, total prostatectomy, cystectomy
* In thoracic surgery: pneumonectomy, lobectomy
* In orthopedic surgery: total hip replacement and total knee prosthesis

Exclusion Criteria:

* pathology making it impossible to measure Systolic Pressure Index
* life expectancy less than 6 months
* emergency surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from thoracic surgery, cardiovascular surgery and transplantation,urologic surgery, gastrointestinal surgery and orthopedic surgery services and coming to a preoperative anesthesia consultation are concerned with the study.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
It is a composite involving the following events: death, cardiovascular death, acute coronary syndrome, left cardiac decompensation, stroke, transient ischemic attack | day1, day 2, day 3, 1 month, 1 year

SECONDARY OUTCOMES:
- for the short term increase in the length of hospitalization - for the long term: death, cardiovascular death, hospitalization for acute coronary syndrome, cardiac decompensation left, TIA, stroke, acute ischemia and ischemia critical member. | day1, day 2, day 3, 1 month, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe LACROIX, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Explorations fonctionnelles vasculaires et angiologie (Hôpital Dupuytren), Limoges, France